CLINICAL TRIAL: NCT03601364
Title: The Effect of PEEP and Tidal Volume on Thiol / Disulphide and Other Oxidative Stress Parameters in Cardio Pulmonary Bypass Surgery
Brief Title: The Effects of Peep and Tidal Volume on Oxidative Stress in Cardiopulmonary Bypass Surgery
Status: Completed | Type: Observational
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Yavuz Orak, Assistant Professor, Kahramanmaras Sutcu Imam University
Other Study IDs: 2018/10-12
Record Dates: First submitted 2018-07-17; First posted 2018-07-26 (Actual); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Cardiac Surgery; Oxidative Stress
Keywords: peep, tidal volume, cardiopulmonary bypass, oxidative stress

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: 1.Mechanical ventilator closed group (Mechanical ventilator off)
- Group 2: 1. Tidal Voltage 3-4ml / kg (TV),
  2. FIO2 50%, Flow: 2L / min,
  3. Frequency; 10-12 applied group.
- Group 3: 1. PEEP: 5 cm H2O basınç,
  1. Tidal Voltage 3-4ml / kg (TV),
  2. FIO2 50%, Flow: 2L / min,
  3. Frequency; 10-12 applied group.

SUMMARY:
Although cardio-pulmonary bypass surgery (CPBS) is a routine procedure worldwide, patient morbidity and mortality are still high due to postoperative negative complications.Inflammatory response and systemic oxidative stress have been reported to be directly related to this practice.Mechanisms explaining this condition have been described as being related to several events that occur during the cardiopulmonary bypass (CPBS), where blood is exposed to non-physiological surfaces, surgical trauma, ischemia-reperfusion, and changes in body temperature.In addition, CPB induces atelectasis and affects the structure of the bronchoalveolar tree.Prolongation of atelectasis may facilitate proinflammatory cytokine production by macrophages.One of the most damaging consequences of all these events is the formation of reactive oxygen species (ROS) and radicals originating from various cellular and enzymatic sources such as myocardial cells, activated neutrophils.ROS has toxic effects on cellular structures including lipids, proteins and nucleic acids.Oxidative reaction damages cellular function and may increase perioperative or postoperative complications after CPBS.Total antioxidant status (TAS), total oxidant status (TOS) and oxidative stress index (OSI) reflect the redox balance between oxidation and antioxidation.TAS measurement is an indication of the activity of all antioxidants and TOS is an indicator of ROS.OSI is a measure of the ratio of TOS to TAS and the level of Oxidative Stress (OS).The contribution of various mechanisms to oxidant-antioxidant balance during on-pump coronary artery bypass grafting (ONCABG) has not yet been fully evaluated. The investigator's aim in this study is to investigate the effect of lung protective mechanism (Tidal Volum, PEEP) on oxidative stress parameters such as TAS, TOS, Thiol / Disulphide, Catalase, Glutathione Peroxidase, MDA (Melanil Dialdehyde) in cardio pulmonary bypass surgery

DETAILED DESCRIPTION:
The study will be performed on patients who accept cardiopulmonary by-pass surgery, the conscious openness to participate in the study.Age, sex, body mass index (BMI), smoking habits, diagnosis, additional diseases, drugs used, surgery, intervention, anesthetic agents used in induction and dyspepsia, peroperative supportive treatments, left ventricular ejection fraction, post operative blood and TDP amount CPB (cardiopulmonary bypass) time (min), Cross clamp time (min), cardioplegia amount and type, analgesic name and dose made, duration of operation, name of postoperative and perioperative support treatments , perioperative and post operative intake and urine output,postoperative extubation time, intensive care day of hospitalization, day of hospitalization will be recorded.The study was planned in 3 groups.Group 1 mechanical ventilator closed group (mechanical ventilator off) FiO2; 50%, Flow: 2 L / min. 2 Group Tidal Volume 3-4ml / kg (TV), FIO2 50%, Flow: 2L / min, Frequency; 10-12 applied group. 3. Group Tidal Volume 3-4 ml / kg, PEEP: 5 cm H2O pressure, FIO2 50%, Flow: 2 L / min, Frequency:Planned to be the 10-12 applied group.Pre-operative, operative (After the cross clamp is removed) and postoperative (postoperative 24th hour) blood will be collected from patients participating in the study.Thiol / Disulphide, MDA, TAS, TOS, Catalase and Glutathione Peroxidase will be studied. All patients should be premedicated with 0.1 mg / kg midazolam.Fentanyl (5-8 μg / kg), and rocuronium (0.5 mg / kg) will be used for induction of anesthesia. During anesthesia, 2% sevoflurane will be used.Arterial cannula to be inserted.Central venous catheter and urinary catheter will be placed. 3 - 5 mg / heparin and cardioplegia will be applied.The active clotting time (ACT) will be kept above 400.Heparin 1: to be neutralized with 1.3% of the Protamine.In the postoperative period, all patients will be transferred to the intensive care unit.

ELIGIBILITY:
Inclusion Criteria

* Patients who will be cardiopulmonary by-pass surgery and volunteer to participate in the study will be included in the study.
* Between 18-80 years

Exclusion Criteria:

* Patients requiring acute coronary syndrome and emergency cardiovascular surgery,
* Patients who have had myocardial infarction within the past month
* Recurrent cardiovascular surgery
* Off-pump coronary artery bypass surgery (OPCAB)
* Patients with chronic inflammatory disease (rheumatoid arthritis, malignancy, psoriasis, etc.), autoimmune disease, immunocompromised patients
* Patients with chronic renal failure, liver disease, active infection
* Patients older than 80 years and smaller than 18 years

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who will be cardiopulmonary by-pass surgery and volunteer to participate in the study will be included in the study.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-10 (Actual)

PRIMARY OUTCOMES:
Oxidative stress markers | Change from baseline before operation (preoperative),peroperative,24 hours after surgery,
  To evaluate the impact on the circulating levels of Catalase ü/ml,Glutathione Peroxidase ü/ml, Malondialdehyde nmol/ ml, Thiol Disulfide,TAS, TOS

SECONDARY OUTCOMES:
supportive care | used during surgery and during the first 24 hours after surgery
  Dopamine, Dobutamine,Gliserol Trinitrat, Adrenalin, Noradrenaline levels
blood and fresh frozen plasma (FFP) | used during surgery and during the first 24 hours after surgery
  blood and fresh frozen plasma (FFP) quantities

CONTACTS AND LOCATIONS:
Overall Officials: yavuz orak, md, Principal Investigator — Kahramanmaraş Sutcu Imam University Faculty of Medicine
Locations (1):
- Kahramanmaras Sutcu Imam University Faculty of Medicine, Kahramanmaraş, Onikişubat, Turkey (Türkiye)